CLINICAL TRIAL: NCT01524315
Title: Preoperative Parenteral Thiamine Supplementation in Patients Undergoing Heart Surgery - a Pilot Study
Brief Title: Preoperative Parenteral Thiamine Supplementation in Patients Undergoing Heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael J. Hiesmayr, Michael Hiesmayr, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2011-004080-70; 2011-004080-70 (EudraCT Number)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure; Acidosis, Lactic; Thiamine Deficiency
Keywords: Thiamine; Vitamin B1; Thiamine Deficiency; Thiamine supplementation; Cardiac surgery; Lactic Acid
MeSH Terms: conditions — Heart Failure; Acidosis, Lactic; Thiamine Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supplementation (Experimental): 6 ml Vitamin-B1-ratiopharm in 100 ml normal saline, intravenous, preoperative
  Interventions: Drug: Vitamin B1-ratiopharm
- Placebo (Placebo Comparator): 100 ml normal saline, intravenous, preoperative
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin B1-ratiopharm — 300 mg Thiaminchloridhydrochlorid, once, intravenous, preoperative
  Other Names: Vitamin B1-ratiopharm®
  Arms: Supplementation
Drug: Placebo — 100 ml normal saline, intravenous, preoperative
  Arms: Placebo

SUMMARY:
The objective of this study is to determine whether preoperative parenteral thiamin supplementation does prevent the intra and early postoperative increase of lactate and whether this effect is related to the extent of thiamine deficiency in patients undergoing heart surgery. In addition the prevalence of major thiamin deficiency in patient undergoing heart surgery will be determined.

DETAILED DESCRIPTION:
Thiamine (vitamin B1) is a water-soluble vitamin and is involved in several stages of intermediate metabolism which are important for producing energy. Severe thiamin deficiency has been associated with severe lactic acidosis and clinical symptoms of life threatening heart failure.

To date, no study has evaluated thiamine levels in patients undergoing heart surgery and the prevalence of thiamine deficiency is not known. Furthermore it is unknown whether moderately reduced thiamin levels are associated with mild forms of perioperative cardiac failure necessitating prolonged inotropic support.

In this prospective double blind randomised controlled trial of the effect of a parenteral infusion of thiamin before induction of anaesthesia we will investigate the effect on perioperative lactate increase as primary outcome and extent and duration of inotropic support after cardiac surgery. In addition the pharmacokinetics of a intravenous infusion of 300 mg of thiamin on erythrocyte thiamin content and the amount of thiamine excreted in the 24 hours via the urine will be determined.

Baseline thiamin levels in erythrocytes before surgery, as well as nutrition history and body composition will be evaluated as effect modifier.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 100 years
* planned heart surgery
* signed informed consent

Exclusion Criteria:

* pregnancy and lactation
* known allergic reaction to the drugs used
* mental condition rendering the patient unable to give informed consent
* inability or contraindications to perform study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-02-02 (Actual)

PRIMARY OUTCOMES:
Thiamine status and lactate levels | perioperative
  Thiamine status: functional parameter - erythrocyte transketolase (α-ETK) expressed as TPP (thiamine pyrophosphate); quantity of vitamin B1 in urine and blood concentrations Lactate levels: lactate levels will be determined by blood gas analysis (BGA) within the routine check.

SECONDARY OUTCOMES:
Prevalence of thiamine deficiency, identification of body composition and length of hospital and ICU stay | 2-3 weeks
  Thiamine status: functional parameter - erythrocyte transketolase (α-ETK) expressed as TPP (thiamine pyrophosphate); Body composition: measuring with bioelectrical impedance analysis (BIA) Length of ICU and hospital stay;

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hiesmayr, Prof.,MD, Principal Investigator — MU Vienna
Locations (1):
- Medical University Vienna, Vienna, Austria

REFERENCES:
- [Result] Luger M, Hiesmayr M, Koppel P, Sima B, Ranz I, Weiss C, Konig J, Luger E, Kruschitz R, Ludvik B, Schindler K. Influence of intravenous thiamine supplementation on blood lactate concentration prior to cardiac surgery: A double-blinded, randomised controlled pilot study. Eur J Anaesthesiol. 2015 Aug;32(8):543-8. doi: 10.1097/EJA.0000000000000205. PMID 26066773